CLINICAL TRIAL: NCT01772875
Title: Pilot Study to Evaluate the Efficacy of Antiseptic Bladder Lavage Versus Pulsatile Lavage With Physiologic Serum in Catheterized Patients With Asymptomatic Bacteriuria With Uropathogens.
Brief Title: Bladder Lavage as Decontamination Method for Asymptomatic Bacteriuria With Uropathogens in Catheterized Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no clinical investigator present
Sponsor: National Multiple Sclerosis Center (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Daphne Kos, Scientific Research, National Multiple Sclerosis Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BLLAV-1
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Catheter Related Infections
Keywords: urinary catheter; UTI; bladder lavage
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- lavage Isobetadine Dermicum solution (Active Comparator): Patient will receive 1 bladder lavage daily with a solution of 5ml Isobetadine Dermicum in 100cc saline
  Interventions: Procedure: bladder lavage
- lavage Acetic Acid solution (Active Comparator): Patients will receive a daily bladder lavage during 5 consecutive days with a solution of 0.5% acetic acid in 100cc of saline
  Interventions: Procedure: bladder lavage
- lavage with saline (Sham Comparator): patients will receive during 5 consecutive days a bladder lavage with 100cc saline
  Interventions: Procedure: bladder lavage
- lavage Urotainer Suby G (Active Comparator): patients will receive during 5 consecutive days a bladder lavage with 100cc of Urotainer Suby G
  Interventions: Procedure: bladder lavage

INTERVENTIONS:
Procedure: bladder lavage — the bladder is rinced through the urinary catheter with the lavage solution
  Other Names: bladder rincing

SUMMARY:
In patients with advanced multiple sclerosis, permanent urinary catheters are often used to manage the urinary incontinence and bladder emptying problems. These catheters will lead to urinary tract infection, blocking of the catheter etc.. Especially infections with certain bacteria such as proteus, enterobacteriaceae and ESBL producing enterobacteriaceae and pseudomonas can pose a problem for the hospital infection control and for the patient.

This study wants to evaluate the potential role of regular bladder lavage with saline, a solution of betadine, an acid solution of acetic acid and of URotainer Twin Suby G ( Braun)in the decontamination of these bladders and the prevention of clinically relevant urinary tract infections.

DETAILED DESCRIPTION:
PAtients will be selected from the catheterised patient population of the National MS Center in Belgium for this prospective randomised comparative pilot studyon bladder lavage.

The potential benefit for the patient is a reduction in number of clinical urinary tract infections and a reduction of antibiotic use.

According to the type of bacteria that is cultured from the urine, patients will be allocated to one of 4 subgroups:

* 30 patients will recieve bladder lavage with a Isobetadine Dermicum Solution
* 20 patients will revieve bladder lavage with acetic acid solutions
* 10 patients will recieve bladder lavage with saline
* 10 patients will receive bladder lavage with Urotainer Suby G

The effect will be measured by two repeat urine cultures after the bladder lavage( 2days and 5 days).

From a safety perspective and to assess the irritation caused by the lavage, white blood cell counts in the urine will be done.

Adverse events will be monitored according to GCP regulations.

ELIGIBILITY:
Inclusion Criteria:

* patients with an indwelling catheter
* catheter associated bacteriuria with proteus, enterobacteriaceae or pseudomonas
* willing and able to give informed consent to the study

Exclusion Criteria:

* patients with a clinically relevant UTI ( fever, pain or cloudy urine)
* cognitively impaired patients
* patients not able or willing to give informed consent
* patients with allergies for ISobetadine dermicum or other substances used in the protocol
* patients who only have a catheter for less than 1 month
* patients taking systemic antibiotics during the last 48h

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01 (Estimated); Primary Completion 2013-12 (Estimated); Study Completion 2014-01-20 (Actual)

PRIMARY OUTCOMES:
urinary culture | day 2 and day 5 after last bladder lavage
  After 5 consecutive days of bladder lavage, a urine culture will be taken at day 2 and 5. A count of <100.000 CFU/ml and is considered a positive result.
  The outcome will be considered positive if this positive result is found in more than 30% of subjects.

SECONDARY OUTCOMES:
pyuria | day 2 and day 5 after the last bladder lavage
  changes in white blood cell count are monitored at day 2 and 5 afte 5 consecutive days of bladder lavage. This is an assessment of bladder irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk De Ridder, Prof., Principal Investigator — National MS Center Belgium & University Hospitals KU Leuven
Locations (1):
- National MS Center, Steenokkerzeel, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Jaggi N, Sissodia P. Multimodal supervision programme to reduce catheter associated urinary tract infections and its analysis to enable focus on labour and cost effective infection control measures in a tertiary care hospital in India. J Clin Diagn Res. 2012 Oct;6(8):1372-6. doi: 10.7860/JCDR/2012/4229.2362. PMID 23205350
- See also: website of the National MS Center, Belgium — http://www.mscenter.be